CLINICAL TRIAL: NCT01860781
Title: The Effect of Paliperidone Palmitate in Schizophrenia: A Prospective Naturalistic Case Series Study
Brief Title: The Effect of Paliperidone Palmitate in Schizophrenia
Acronym: sustenna
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Yong Min Ahn, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R092670-SCH-4008
Record Dates: First submitted 2013-05-21; First posted 2013-05-23 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Injection; Switch; Paliperidone; refractory, chronic akathisia, poor complianc
MeSH Terms: conditions — Schizophrenia | interventions — Paliperidone Palmitate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- paliperidone palmitate (Experimental): paliperidone palmitate
  Interventions: Drug: paliperidone palmitate

INTERVENTIONS:
Drug: paliperidone palmitate — paliperidone palmitate 150mgeq(1 day), 100mgeq(8days), 75mg(monthly)
  Other Names: paliperidone palmitate(sustenna)

SUMMARY:
The purpose of this study is the evaluation of effectiveness of paliperidone palmitate within three different group of schizophrenia patients.

DETAILED DESCRIPTION:
In this study, the investigators are going to examine the effectiveness of paliperidone palmitate after changing from other antipsychotics. This study design is a Prospective Naturalistic Case Series Study. The effectiveness of paliperidone would be compared within three different groups of schizophrenia. Investigators would also assess the safety during 24 weeks follow up period.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 ~ 65
* Patient with schizophrenia according to DSM-IV criteria
* Patient have signed on the informed consent, and well understood the objective and procedure of this study.
* PANSSS total score <120
* each Score of disorganized thought, paranoia hallucinatory behavior, abnormal tbought contests < 16
* three different groups ( other antipsychotics refractory schizophrenia patitents : CGI> 4 chronic akathisia : DIEPSS overall severity >1, at least 1 month lasting symptoms poor compliance schizophrenia : CRS <3)
* Competent patient who is manage to answer the questionnaires.
* In case of female at child-bearing age, consent to use appropriate contraceptive methods(oral pill, contraceptive injection, intrauterine device, double barrier method and contraceptive patch) during entire duration of this study.

Exclusion Criteria:

* No history of antipsychotics prescription
* History of NMS(Neuroleptic malignant syndrome)
* Allergic reaction or hypersensitive reaction of risperidone or paliperidone ER
* clozapine medication within 1 month before screening
* SSRI, MAOI, TCA medication within 2 months
* Lithium, valproic acid, carbamazepine, topiramate, lamotrigine medication starting within 2 months
* patient who is supposed to be impossible to participate to this study due to clinical risk of suicide or aggressive behavior based on clinician's opinion
* current or previous history of drug depedence according to DSM-IV
* Pregnant or breast-feeding female patient
* Significant biochemical or hematological abnormality or abnormal finding of urinalysis, based on clinician's opinion
* history of cardiac disease, which is related to QT prolongation(sick sinus, complete AV block, CHF, ventricular tachycardia, hypokalemia or hypocalcemia)
* History of participating to other investigational drug trial within 1month prior to screening
* Investigator or employee at clinical trial center, personnel related to investigator or trial center on this or other study, or family of employee or investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
CGI-S,I: Clinical Global Impression-Severity, Improvement | 24 weeks

SECONDARY OUTCOMES:
PANSS: Positive and Negative Syndrome Scale | 24 weeks
CRS: Clinician Rating Scale | 24 weeks
KDAI-10: Korean Drug Attitude Inventory-10 | 24 weeks
SWN: Subjective Well-being Under Neuroleptic Treatment | 24 weeks
DIEPSS: Drug-Induced ExtraPyramidal Symptoms Sclae | 24 weeks
injection site pain -VAS: Visual Analog Scale | 24 weeks
LUNSERS: Liverpool University Neuroleptic Side Effect Rating Scale | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Yong Min Ahn, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea